CLINICAL TRIAL: NCT01019707
Title: A Study to Assess the Cardiovascular, Cognitive and Subjective Effects of Atomoxetine in Combination With Intravenous Methamphetamine
Brief Title: Safety Assessment of Atomoxetine With MA IV Administration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: End in funding
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50-18185-PI-EDL-A; P50DA018185 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Methamphetamine Abuse; Methamphetamine Dependence
Keywords: crystal meth; methamphetamine; substance abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): As this is a within-subject, crossover design, all subjects complete both study medication assignments in a double-blind fashion. Based on random assignment to start on either atomoxetine or placebo, study drug will be administered once daily at 40 mg/day on the first 2 study days, then twice daily for the third, fourth and fifth study days, and once daily on the sixth study day.
  Interventions: Drug: Atomoxetine, then Placebo; Drug: Placebo, then Atomoxetine
- Atomoxetine (Active Comparator): As this is a within-subject, crossover design, all subjects complete both study medication assignments in a double-blind fashion. Based on random assignment to start on either atomoxetine or placebo, study drug will be administered once daily at 40 mg/day on the first 2 study days, then twice daily for the third, fourth and fifth study days, and once daily on the sixth study day.
  Interventions: Drug: Atomoxetine, then Placebo; Drug: Placebo, then Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine, then Placebo — As this is a within-subject, crossover design, all subjects complete both study medication assignments in a double-blind fashion. Based on random assignment to start on either atomoxetine or placebo, study drug will be administered once daily at 40 mg/day on the first 2 study days, then twice daily for the third, fourth and fifth study days, and once daily on the sixth study day.
  Other Names: Strattera
Drug: Placebo, then Atomoxetine — As this is a within-subject, crossover design, all subjects complete both study medication assignments in a double-blind fashion. Based on random assignment to start on either atomoxetine or placebo, study drug will be administered once daily at 40 mg/day on the first 2 study days, then twice daily for the third, fourth and fifth study days, and once daily on the sixth study day.

SUMMARY:
This is a study of 4 nontreatment seeking individuals who were MA-dependent and the safety and tolerability of atomoxetine. This double-blind, placebo-controlled, within-subjects study is to determine the safety and tolerability of atomoxetine.

MA abusing participants will undergo a 1-day outpatient screening and if it is safe for the participants to proceed with the study they will participate in two inpatient components of the study that will occur in the University of California Los Angeles (UCLA) General Clinical Research Center (GCRC). The first inpatient stay will be 15 days, and the second will be a 9 days stay that includes drug administration and assessments. There will be at least a two week interval between inpatient components. During the inpatient components participants will receive alternating study drugs; atomoxetine or placebo and four sessions of IV MA administration or saline.

DETAILED DESCRIPTION:
The safety of using atomoxetine in MA users will be characterized by measuring the cardiovascular effects of MA and by determining the occurrence of adverse reactions during treatment with atomoxetine and placebo. We will evaluate atomoxetine (0 and 40 mg, BID) and MA doses (0 and 30 mg, IV).

Participants will be randomized to atomoxetine or matched placebo for 6 days. Study drug will be administered once daily at 40 mg/day on the first two study days, twice daily for days 3-5, & once on day 6. After discharge from the first component, and at least a 2-week washout period, participants will be re-admitted to the UCLA GCRC and switched to the opposite study medication for an additional 6 days.

Methamphetamine/saline will be administered non-contingently on component I day 13, and component II day 7, over 1 min using a syringe pump activated by the study physician or nurse practitioner in order to assess safety and tolerability of atomoxetine. During drug administration sessions, heart rate and blood pressure will be monitored frequently. A code team will respond if required. Vital signs must remain within values specified under Stopping Criteria for initiation of MA administration. The physician or nurse practitioner will administer the MA/placebo and will be available in-house on pager for at least 4 h after each infusion. In addition, heart rate and blood pressure will be assessed three times daily throughout the inpatient portion of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Be fluently English-speaking volunteers who meet DSM-IV criteria for MA abuse or dependence.
2. Be between 18 and 50 years of age.
3. Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
4. Have smoked or injected methamphetamine for more than two years.
5. Produce a methamphetamine-positive urine prior to study entry.
6. Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 105-150mm Hg systolic and 45-90mm Hg diastolic. Note that a blood pressure of 150/90 and pulse of 90 is too high for randomization but will allow participants to be enrolled if an acceptable range is demonstrated on a separate occasion.
7. Have an ECG performed that demonstrates normal sinus rhythm, normal conduction, and no clinically significant arrhythmias.
8. Agree to abstain from MA during the study, evidenced by a MA-negative urine each morning of the study.
9. If female, have a negative pregnancy test and agree to use one of the following methods of birth control, or be postmenopausal, have had a hysterectomy or have been sterilized.

   1. oral contraceptives
   2. barrier (diaphragm or condom) with spermicide, or condom only
   3. intrauterine progesterone,or non-hormonal contraceptive system
   4. levonorgestrel implant
   5. medroxyprogesterone acetate contraceptive injection
   6. complete abstinence from sexual intercourse

NOTE: Recent intermittent alcohol or other illicit drug use without physical dependence is allowable (however a benzodiazepine-free urine should be produced to document absence of recent use).

Exclusion Criteria:

1. A current or past history of seizure disorder, including alcohol- or stimulant-related seizure, febrile seizure, or significant family history of idiopathic seizure disorder.
2. A history of head trauma that resulted in neurological sequelae (e.g., with loss of consciousness [LOC] > 15 minutes, or that required hospitalization. Also, individuals with 3 or more head injuries with LOC > 5 minutes will be excluded).
3. Do not meet DSM-IV criteria (by SCID) for drug dependence other than meth, with the exception of nicotine and/or marijuana dependence.
4. Any previous medically serious adverse reaction to MA including loss of consciousness, chest pain, or epileptic seizure resulting in hospitalization.
5. Meeting diagnostic criteria or receiving psychopharmacological treatment for the following Axis I disorders within the last 6 months: anorexia nervosa, bulimia, psychosis, bipolar I disorder, organic brain disease, dementia, major depression, schizoaffective disorder, or schizophrenia.
6. Evidence of clinically significant heart disease, hypertension or significant medical illness.
7. Have any history of hypersensitivity to atomoxetine, glaucoma, motor tics or with a family history or diagnosis of Tourette's syndrome.
8. Have any preexisting severe gastrointestinal narrowing, small bowel inflammatory disease, intestinal adhesions, past history of peritonitis, or cystic fibrosis.
9. Be pregnant or nursing.
10. Have a significant family history of early cardiovascular morbidity or mortality.
11. Have a diagnosis of adult asthma, including those with a history of acute asthma within the past two years, and those with current or recent (past 2 years) treatment with inhaled or oral beta-agonist or steroid therapy (due to potential serious adverse interactions with methamphetamine).
12. Be actively using albuterol or other beta agonist medications, regardless of formal diagnosis of asthma. (Inhalers are sometimes used by MA addicts to enhance MA delivery to the lungs.) If respiratory disease is excluded and the subject will consent to discontinue agonist use, s/he may be considered for inclusion.
13. For subjects suspect for asthma but without formal diagnosis, 1) have a history of coughing and/or wheezing, 2) have a history of asthma and/or asthma treatment two or more years before, 3) have a history of other respiratory illness, e.g., complications of pulmonary disease (exclude if on beta agonists), 4) use over-the-counter agonist or allergy medication for respiratory problems (e.g., Primatene Mist): a detailed history and physical exam, pulmonary consult, and pulmonary function tests should be performed prior to including or excluding from the study or 5) have an FEV1 <70 %.
14. Have any illness, condition, and/or use of medications that in the opinion of the site Principal Investigator and the admitting physician would preclude safe and/or successful completion of the study.
15. Have active syphilis that has not been treated or refuse treatment for syphilis.
16. Be undergoing HIV treatment with antiviral and non-antiviral therapy.
17. Have AIDS according to the current CDC criteria for AIDS - MMWR 1999;48 (#RR-13:29-31).
18. Have neurological disorders including Parkinson's disease.
19. Have evidence of significant liver or kidney dysfunction.
20. Have a history of urinary retention or bladder outlet obstruction.
21. Be UCLA students or staff.
22. Have evidence of active tuberculosis infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoptaw, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute NPI, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects will be self-identified as non-treatment seeking MA users recruited via advertisements in online sources and newspapers, on radio stations, and community locations, as well as through referrals from within as well as from outside organizations via flyers, and from past research participants.
Pre-assignment Details: MA-dependent, non-treatment seeking subjects only were enrolled in this study. A screening period to assess eligibility criteria was used to determine study eligibility. Study completion involved finishing a 15-day inpatient period,followed by 14+ days washout in community, followed by a second 9-day inpatient period.
Groups:
- Atomoxetine, Then Placebo: In this double-blind, within-subject crossover clinical trial, subjects received MA infusion and saline infusions under atomoxetine for 15 days and then placebo for 9 days after a 14 day wash out. The order of study drug was determined randomly.
- Placebo, Then Atomoxetine: In this double-blind, within-subject crossover clinical trial, subjects received MA infusion and saline infusions under placebo for 15 days and then atomoxetine for 9 days after a 14 day wash out. The order of study drug was determined randomly.
Period: First Phase
Arm/Group | Atomoxetine, Then Placebo | Placebo, Then Atomoxetine
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Washout
Arm/Group | Atomoxetine, Then Placebo | Placebo, Then Atomoxetine
Started | 3 | 3
Completed | 3 | 1
Not Completed | 0 | 2
Period: Second Phase
Arm/Group | Atomoxetine, Then Placebo | Placebo, Then Atomoxetine
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Four (4) subjects completed both components (atomoxetine and placebo) in this double-blind, placebo-controlled crossover trial design.
Groups:
- Total Sample: In this double-blind, within-subject crossover clinical trial, subjects received MA infusion and saline infusions under atomoxetine and placebo. The order of study drug was determined randomly.
Arm/Group | Total Sample
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Based on 8 timepoints post MA infusion, data were pooled and the mean value and standard deviation are presented. Timepoints assessed were collected at 2, 5, 10, 15, 30, 45, 60, 90 minutes following infusion.
Time Frame: Timepoints post MA infusion
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: Timepoints
Groups:
- Atomoxetine With MA; Placebo With MA: Based on random assignment, study drug will be administered once daily at 40 mg/day on the first 2 study days, then twice daily for the third, fourth and fifth study days, and once daily on the sixth study day. Subjects received up to 30mg MA during one study day per medication condition.
Arm/Group | Atomoxetine With MA | Placebo With MA
Number analyzed (Participants) | 4 | 4
Number analyzed (Timepoints) | 32 | 32
mm Hg | 126.2 (15.3) | 137.1 (14.7)

2. Primary Outcome: Diastolic Blood Pressure
Description: as for outcome 1
Time Frame: Timepoints post MA infusion
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: Timepoints post infusion
Arm/Group | Atomoxetine With MA | Placebo With MA
Number analyzed (Participants) | 4 | 4
Number analyzed (Timepoints post infusion) | 32 | 32
mm Hg | 72.4 (10.6) | 79.3 (13.5)

3. Primary Outcome: Heart Rate
Description: as for outcome 1
Time Frame: Timepoints post MA infusion
Measure: Mean (Standard Deviation); unit: BPM
Units Other Than Participants: Timepoints
Arm/Group | Atomoxetine With MA | Placebo With MA
Number analyzed (Participants) | 4 | 4
Number analyzed (Timepoints) | 32 | 32
BPM | 81.3 (15.3) | 82.1 (13.2)

ADVERSE EVENTS:
Groups:
- Atomoxetine With MA; Placebo With MA: Based on random assignment, study drug will be administered once daily at 40 mg/day on the first 2 study days, then twice daily for the third, fourth and fifth study days, and once daily on the sixth study day. Subjects received infusions of saline and 30mg MA on one study day per medication condition.
Arm/Group | Atomoxetine With MA | Placebo With MA
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine With MA (N=4) | Placebo With MA (N=4)
Headache (General disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 2 (2) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subject analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes